CLINICAL TRIAL: NCT00992186
Title: An Open-Label, Multicenter, Phase 2 Study of Single-Agent CNTO 888 (an Anti-CCL2 Monoclonal Antibody) for the Treatment of Subjects With Metastatic Castrate-Resistant Prostate Cancer
Brief Title: A Study of the Safety and Efficacy of Single-agent Carlumab (an Anti-Chemokine Ligand 2 [CCL2]) in Participants With Metastatic Castrate-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centocor Research & Development, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015907; 2009-011251-48; CNTO888PCR2001
Record Dates: First submitted 2009-09-29; First posted 2009-10-09 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Infusion; Carlumab; CNTO 888
MeSH Terms: conditions — Prostatic Neoplasms | interventions — carlumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carlumab (Experimental)
  Interventions: Drug: Carlumab

INTERVENTIONS:
Drug: Carlumab — Carlumab diluted in 5 percent (%) dextrose administered at the dose of 15 milligram per kilogram (mg/kg) by intravenous (into a vein) infusion (a fluid or a medicine delivered into a vein by way of a needle) at a constant rate over a 90 minute period once every 2 weeks until disease progression.

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of the study drug carlumab in participants with metastatic castrate-resistant prostate cancer (cancer of the gland that makes fluid that aids movement of sperm).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multicenter trial (conducted in more than one center) in participants with metastatic castrate-resistant prostate cancer. The trial consists of 3 phases: screening period, treatment period of approximately 4 months, and a follow-up period (Week 1, 4, 8 and 12 after the last dose) of up to 12 weeks after the administration of last dose. The participants will receive carlumab at the dose of 15 milligram/kilogram (mg/kg) by intravenous (into a vein) infusion (a fluid or a medicine delivered into a vein by way of a needle) at a constant rate over a 90 minute period once every 2 weeks until disease progression. Efficacy of the participants will be primarily evaluated by composite response. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histological documentation of adenocarcinoma of the prostate
* Received at least 1 but no more than 2 prior docetaxel-based chemotherapy regimens and had disease progression following the last therapy
* Serum prostate specific antigen (PSA) greater than or equal to 5.0 nanogram/milliliter (ng/ml) within 4 weeks prior to the first dose of study agent
* Orchiectomy (surgery to remove one or both testicles) or testosterone less than 50 nanogram/deciliter by means of pharmacological/chemical castration within 4 weeks prior to the first dose of study agent
* At least 6 weeks from prior docetaxel chemotherapy regimen to first dose of study agent

Exclusion Criteria:

* Experience a hormonal treatment withdrawal response (including a lowering of PSA that was previously rising or symptomatic improvement)
* Known or symptomatic Central Nervous System metastases
* Residual toxicities resulting from previous therapy that are Grade 2 or more (except for alopecia)
* Known allergies, hypersensitivity, or intolerance to carlumab or its excipients or clinically significant reactions to chimeric or human proteins
* Vaccinated with live, attenuated vaccines within 4 weeks prior to the first dose of study agent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor Research & Development, Inc., PA, USA Clinical Trial, Study Director — Centocor Research & Development, Inc.
Locations (13):
- United States (3):
  - Orange City, Florida
  - Ann Arbor, Michigan
  - Charleston, South Carolina
- Belgium (3):
  - Antwerp
  - Brussels
  - Wilrijk
- Russia (2):
  - Moscow
  - Saint Petersburg
- United Kingdom (5):
  - Birmingham
  - Guildford
  - Leeds
  - Southampton
  - Sutton

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 out of 62 participants, who signed informed consent, were deemed ineligible for the study during screening because of screening failure, serious adverse events, unavailability of carlumab at the site and withdrawal of consent.
Period: Overall Study
Arm/Group | Carlumab
Started | 46
Completed | 0
Not Completed | 46
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 1
Not completed — Physician Decision | 1
Not completed — Adverse Event | 9
Not completed — Progressive Disease | 30
Not completed — Refusal To Receive Study Agent | 3

BASELINE CHARACTERISTICS:
Arm/Group | Carlumab
Number analyzed (Participants) | 46
Age Continuous [Mean (Standard Deviation); unit: Years] | 67.5 (7.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 46
Region of Enrollment [Number; unit: participants]
  Belgium | 11
  Russian Federation | 10
  United Kingdom | 18
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Composite Response
Description: The composite response is measured by change from Baseline in skeletal lesions, extra-skeletal lesions, and prostate specific antigen (PSA) values. A participant is considered to have composite response, if 1 of the following responses occurs after the first dose of carlumab: (1) Complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST), (2) PSA response at 12 weeks and absence of skeletal and extra-skeletal progression or (3) Stable disease at 24 weeks defined as the absence of PSA, skeletal, or extra-skeletal progression.
Time Frame: Up to 4 weeks before first dose, every 12 weeks after first dose, Week 12 after last dose of carlumab
Population: Analysis population included all the participants who received at least 1 administration of carlumab and had at least 1 post-baseline disease evaluation. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Carlumab
Number analyzed (Participants) | 41
Percentage of participants
  CR or PR | 0.0
  PSA response | 0.0
  Stable disease | 2.4

2. Secondary Outcome: Percentage of Participants With Objective Tumor Response
Description: Objective response based on assessment of confirmed CR or PR according to RECIST. CR defined as disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to less than 10 millimeter (mm). PR defined as at least 30 percent (%) decrease in sum of the diameters of the target lesions taking as reference the Baseline sum diameters. Confirmed responses are those that persist on repeat imaging study for at least 4 weeks after initial documentation of response.
Time Frame: Up to 4 weeks before first dose, every 12 weeks after first dose, Week 12 after last dose of carlumab
Population: Analysis population included all the participants who received at least 1 administration of carlumab and had a measurable, non-measurable or bone lesion at Baseline and had at least 1 post-treatment tumor evaluation. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: Percentage of participants
Groups:
- Carlumab: Carlumab diluted in 5% dextrose administered at the dose of 15 mg/kg by intravenous infusion at a constant rate over a 90 minute period once every 2 weeks until disease progression.
Arm/Group | Carlumab
Number analyzed (Participants) | 41
Percentage of participants
  CR | 0.0
  PR | 0.0

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: The PFS is defined as the time from the date of initiation of study treatment to the date of initial documented skeletal or extra-skeletal progressive disease, or date of death, whichever occurs first. A participant is considered to have extra-skeletal disease progression if the disease has progressed as per the Response Evaluation Criteria in Solid Tumors (RECIST v1.1) criteria. A participant is considered to have skeletal disease progression if they have 1 post-baseline bone scan demonstrating 2 or more new skeletal lesions compared to Baseline and confirmed by a second bone scan 6 to 12 weeks later or with evidence of clinical progression.
Time Frame: Up to 4 weeks before first dose, every 12 weeks after first dose, Week 12 after last dose of carlumab
Population: Analysis population included all the participants who received at least 1 administration of carlumab.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Carlumab
Number analyzed (Participants) | 46
Days | 81.0 [76.0 to 85.0]

4. Secondary Outcome: Overall Survival (OS)
Description: The OS is defined as the time from the date of initiation of study treatment to death due to any cause. Participants were followed for 1 year after the last administration of carlumab for survival or until the end of study, whichever occurs first. For participants with unknown survival status as of the data cutoff date, OS was censored at the last date that the participant was known to be alive.
Time Frame: Week 8, 12, every 12 weeks up to 1 year after last dose of carlumab
Population: Analysis population included all the participants who received at least 1 administration of carlumab.
Measure: Median (Full Range); unit: Days
Arm/Group | Carlumab
Number analyzed (Participants) | 46
Days | 309.0 [47 to 582]

5. Secondary Outcome: Percentage of Participants With Prostate Specific Antigen (PSA) Response
Description: The PSA response for participants with elevated PSA levels at Baseline (more than or equal to 5 nanogram per milliliter (ng/mL) is defined as at least a 50% reduction in PSA from the Baseline value, confirmed by a second PSA value measurement 3 or more weeks later.
Time Frame: Up to 2 weeks before first dose, every 4 weeks after first dose, Week 4, 8, 12 after the last dose of carlumab
Population: Analysis population included all the participants who received at least 1 administration of carlumab and had a Baseline PSA more than or equal to 5 ng/mL and at least 1 post-treatment PSA measurement. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Carlumab
Number analyzed (Participants) | 44
Percentage of participants | 0.0

6. Secondary Outcome: Percentage of Participants With Urinary Crosslinked N-Telopeptide of Type I Collagen (NTx) Response
Description: Urinary NTx response for participants with elevated NTx level at Baseline (more than or equal to 50 nanomole per millimole (nmol/mmol)) is defined as a 30% reduction from Baseline NTx value, confirmed by a second NTx value 3 or more weeks later.
Time Frame: Up to 2 weeks before first dose, every 4 weeks after first dose, Week 4, 8, 12 after the last dose of carlumab
Population: Analysis population included all the participants who received at least 1 administration of carlumab and had elevated urinary NTx level at Baseline (more than or equal to 50 nmol/mmol) and at least 1 post-treatment urinary NTx measurement. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Carlumab
Number analyzed (Participants) | 7
Percentage of participants | 0.0

7. Secondary Outcome: Percentage of Participants With Pain Response
Description: Pain response is defined as 2-point decrease from Baseline in 'worst pain' intensity score (item 3) on the Brief Pain Inventory (BPI) questionnaire. The BPI is a nine-item questionnaire with 0 to 10 numeric rating scales in response to each item, where 0=No pain and 10=Pain as bad as you can imagine. Measure can be scored by item, with lower scores being indicative of less pain or pain interference.
Time Frame: Up to 2 weeks before first dose, every 4 weeks after first dose, Week 4 after last dose of carlumab
Population: Analysis population included all the participants who received at least 1 administration of carlumab, had Baseline BPI 'worst pain' intensity score (item 3) more than or equal to 2, and at least 1 post-treatment pain evaluation. Participants with disease progression were considered to be evaluable, regardless of the post-dose evaluation.
Measure: Number; unit: Percentage of participants
Arm/Group | Carlumab
Number analyzed (Participants) | 31
Percentage of participants
  During stable use of analgesic medication | 32.3
  At any time | 38.7

8. Secondary Outcome: Time to Radiologic Response
Description: Radiologic response based on assessment of confirmed CR or PR according to RECIST. CR defined as disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to less than 10 millimeter (mm). PR defined as at least 30% decrease in sum of the diameters of the target lesions taking as reference the Baseline sum diameters. Confirmed responses are those that persist on repeat imaging study for at least 4 weeks after initial documentation of response.
Time Frame: Up to 4 weeks before first dose, every 12 weeks after first dose, Week 12 after last dose of carlumab
Population: Analysis population included all the participants who received at least 1 administration of carlumab. No data was available for this endpoint as no participant achieved CR or PR.
Arm/Group | Carlumab
Number analyzed (Participants) | 0

9. Secondary Outcome: Duration of Radiologic Response
Description: as for outcome 8
Time Frame: Up to 4 weeks before first dose, every 12 weeks after first dose, Week 12 after last dose of carlumab
Population: as for outcome 8
Arm/Group | Carlumab
Number analyzed (Participants) | 0

10. Secondary Outcome: Minimum Observed Serum Concentration (Cmin)
Time Frame: Pre-dose and at the end of infusion for each Dose; 2, 4 hour (hr) and 1 week after Dose 1; 2 hr after Dose 4; Week 1, 4, 8 and 12 post-last dose
Population: Analysis population included all the participants who received at least 1 administration of carlumab. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: microgram/milliliter (mcg/mL)
Arm/Group | Carlumab
Number analyzed (Participants) | 35
microgram/milliliter (mcg/mL) | 91.82 (87.240)

11. Secondary Outcome: Maximum Observed Serum Concentration (Cmax)
Description: The maximum observed analyte concentration was measured.
Time Frame: as for outcome 10
Population: Analysis population included all the participants who received at least 1 administration of carlumab.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Carlumab
Number analyzed (Participants) | 46
mcg/mL | 320.27 (75.712)

12. Secondary Outcome: Area Under the Serum Concentration Versus Time Curve Between 0 And 14 Days (AUC 0-14d)
Time Frame: Pre-dose, at the end of infusion, 2, 4 hr and 1 week after end of infusion for the first dose
Population: Analysis population included all the participants who received at least 1 administration of carlumab except those whose serum samples were missing at the end of infusion.
Measure: Mean (Standard Deviation); unit: mcg*day/mL
Arm/Group | Carlumab
Number analyzed (Participants) | 41
mcg*day/mL | 1635.67 (528.925)

13. Secondary Outcome: Half-life (t1/2)
Description: The time measured for the serum concentration to decrease by one half.
Time Frame: as for outcome 10
Population: as for outcome 12
Measure: Median (Full Range); unit: Days
Arm/Group | Carlumab
Number analyzed (Participants) | 7
Days | 13.32 [8.7 to 20.0]

14. Other Pre Specified Outcome: Time to Worsening in Eastern Cooperative Oncology Group (ECOG) Status Score
Description: A worsening in ECOG performance status score was defined as greater than or equal to 1-point increase from Baseline. Time to worsening is defined as the number of days from first dose to the first day of worsening in ECOG score, or death, whichever occurred first. ECOG is a 5-point scale 0=Fully active, 1=Ambulatory, carry out work of sedentary nature, 2=Ambulatory, capable of all selfcare, 3=Capable of limited selfcare, confined to bed or chair more than 50% of waking hours, 4=Completely disabled, no selfcare, totally confined to bed or chair, 5=Dead.
Time Frame: Up to 2 weeks before first dose, pre-infusion, Week 4 after last dose of carlumab
Population: Analysis population included all the participants who received at least 1 administration of carlumab.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Carlumab
Number analyzed (Participants) | 46
Days | 86.0 [56.0 to 176.0]

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after last dose of carlumab
Arm/Group | Carlumab
Serious Adverse Events (participants affected / at risk) | 20/46
Other Adverse Events (participants affected / at risk) | 40/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carlumab (N=46)
General physical health deterioration (General disorders) | 1
Multi-organ failure (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Spinal cord compression (Nervous system disorders) | 3
Nerve root compression (Nervous system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Vitreous detachment (Eye disorders) | 1
Confusional state (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carlumab (N=46)
Back pain (Musculoskeletal and connective tissue disorders) | 15
Bone pain (Musculoskeletal and connective tissue disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6
Groin pain (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4
Fatigue (General disorders) | 24
Oedema peripheral (General disorders) | 6
Asthenia (General disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 11
Dehydration (Metabolism and nutrition disorders) | 3
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 4
Confusional state (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4
Gastroenteritis (Infections and infestations) | 3
Weight decreased (Investigations) | 3
Hypertension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If Investigator wishes to publish information from study, a copy of manuscript must be provided to Sponsor for review at least 60 days before publication. Expedited reviews will be arranged for abstracts, poster presentations. If requested by Sponsor in writing, Investigator will withhold such publication for up to additional 60 days to allow for patent filing. If the issues arise regarding scientific integrity or regulatory compliance, Sponsor will review them with Investigator.